CLINICAL TRIAL: NCT03532295
Title: Safety and Efficacy Study of Retifanlimab and Epacadostat in Combination With Radiation and Bevacizumab in Patients With Recurrent Gliomas
Brief Title: Retifanlimab and Epacadostat in Combination With Radiation and Bevacizumab in Patients With Recurrent Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202003050
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — epacadostat; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Regimen A: Retifanlimab+RT+bevacizumab (Experimental): * Retifanlimab will be given intravenously over the course of 30 to 60 minutes at a dose of 500 mg on Day 1 of each 28-day cycle.
  * Bevacizumab will be given intravenously at a dose of 10 mg/kg on Days 1 and 15 of each 28-day cycle.
  * Ten fractions of radiation therapy will be given at a dose of 3.5 Gy per fraction
  * Retifanlimab and bevacizumab will be started approximately two weeks before the first day of radiation therapy
  * Treatment may continue for up to two years.
  Interventions: Drug: Bevacizumab; Radiation: Radiation therapy; Drug: Retifanlimab
- Regimen B: Retifanlimab+RT+bevacizumab+epacadostat (Experimental): * Retifanlimab will be given intravenously over the course of 30 to 60 minutes at a dose of 500 mg on Day 1 of each 28-day cycle.
  * Bevacizumab will be given intravenously at a dose of 10 mg/kg on Days 1 and 15 of each 28-day cycle.
  * Ten fractions of radiation therapy will be given at a dose of 3.5 Gy per fraction
  * Retifanlimab and bevacizumab will be started approximately two weeks before the first day of radiation therapy
  * Epacadostat will be administered orally at 400 mg BID.
  * Treatment may continue for up to two years.
  Interventions: Drug: Epacadostat; Drug: Bevacizumab; Radiation: Radiation therapy; Drug: Retifanlimab

INTERVENTIONS:
Drug: Epacadostat — -All BID doses will be taken in the morning and evening, approximately 12 hours apart
  Arms: Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Drug: Bevacizumab — -The first infusion will be over the course of 90 minutes; if tolerated, the second infusion will be over the course of 60 minutes; if tolerated, all subsequent infusions will be over 30 minutes
  Other Names: Avastin
Radiation: Radiation therapy — -The gross tumor maximum diameter (to be irradiated) to be </= 6 cm in the first 6 patients. If more than 1 target is irradiated, then the sum of all the target maximum diameters should be </= 6 cm. No more than 3 separate targets for RT is allowed.
Drug: Retifanlimab — -Will be supplied by Incyte
  Other Names: INCMGA00012

SUMMARY:
In this study, the investigators propose to combine retifanlimab with radiation therapy (RT) and bevacizumab with or without epacadostat in the treatment of recurrent glioblastoma (GBM). The investigators hypothesize that this combination provides a powerful synergy between RT and immune modulators to produce more robust anti-tumor immune response, induce tumor regression and improve overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent WHO grade 4 glioblastoma or gliosarcoma, including molecular features of glioblastoma and WHO grade 4 astrocytoma or WHO grade high grade glioma.
* Other GBM variants and "secondary GBM" are allowed. All grade 4 gliomas that have relapsed more than once may be included, as the prognosis of multiply recurrent grade 4 glioma patients may not differ based on IDH mutation status.
* Disease must have recurred, and patient must be a candidate for re-irradiation and bevacizumab. Any number of recurrences are allowed.
* Patients must have measurable disease per RANO criteria. Lesions will be considered measurable when they are bi-dimensional with clearly defined margins of ≥5 mm in two perpendicular diameters.
* Prior transient use of bevacizumab for cerebral edema or radiation necrosis is allowed without a washout period. Prior bevacizumab use is permitted if used for treatment of disease if administered more than 4 months prior to registration.
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 9.0 g/dL or > 5.6 mmol/L (transfusion is acceptable to meet this criterion)
  * Serum creatinine ≤ ULN or creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault for patients
  * Serum total bilirubin ≤ 1.5 ULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * INR or PT ≤ 1.5 x IULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* At least 28 days from any major surgery such as craniotomy and surgical wound is fully healed, and at least 14 days from LITT or biopsy. Prior to surgery, there must be imaging evidence of measurable progressive disease (PD) per RANO criteria as noted above.
* Women of childbearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Prior use of the Optune device is allowed, without a washout period. However, concurrent Optune use is not permitted while on treatment for this trial.

Exclusion Criteria:

* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to epacadostat, retifanlimab, bevacizumab, or other agents used in the study.
* Dexamethasone dose > 4 mg daily at the time of registration (higher dose of steroid for symptom control is allowed during the study).
* History of intracranial abscess within 6 months prior to start of study therapy.
* Has active autoimmune disease or syndrome (i.e. moderate or severe rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, active inflammatory bowel disease) that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) or who are receiving systemic therapy for an autoimmune or inflammatory disease (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Subjects are permitted to enroll if they have vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Has a severe acute or chronic medical condition including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Has had an allogeneic tissue/solid organ transplant.
* Has an active infection requiring intravenous antibiotic therapy. Has a known history of active tuberculosis (TB; bacillus tuberculosis).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or IDO inhibitor.
* If a patient is enrolled to regimen B, they are prohibited from receiving monoamine oxidase inhibitors (MAOIs) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.
* If a patient is enrolled to regimen B, the use of any UGT1A9 inhibitor from screening through follow-up period, including acitretin, amitriptyline, androsterone, cyclosporine, dasatinib, diclofenac, diflunisal, efavirenz, erlotinib, estradiol (17-beta), flutamide, gefitinib, gemfibrozil, glycyrrhetinic acid, glycyrrhizin, imatinib, imipramine, ketoconazole, linoleic acid supplements, mefenamic acid, mycophenolic acid, niflumic acid, nilotinib, phenobarbital, phenylbutazone, phenytoin, probenecid, propofol, quinidine, ritonavir, sorafenib, sulfinpyrazone, valproic acid, and verapamil is prohibited.
* If a patient is enrolled to regimen B, the use of probiotics from screening through end of treatment is prohibited.
* If a patient is enrolled to regimen B, the use of warfarin is prohibited. If anti-coagulation is needed during the conduct of the study and non-warfarin regimens are not feasible, the participant must discontinue study therapy.
* Chronic use of systemic antibiotics (> 14 days) unless medical monitor review and approval.
* Any history of serotonin syndrome (SS) after receiving serotonergic drugs.
* Has uncontrolled HIV (HIV 1/2 antibodies). Well-controlled HIV is defined as CD4+ count > 300 cells, undetectable viral load, and receiving HAART/ART. Study specific HIV testing is not required for patients who do not have any prior history of HIV.
* Has uncontrolled active hepatitis B (e.g., HBsAg reactive or HBV DNA detected by quant RT PCR) or hepatitis C (e.g. HCsAg reactive or HCV RNA [qualitative or quantitative] is detected).
* Uncontrolled intercurrent illness including, but not limited to, clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 60 months prior to enrollment), congestive heart failure (≥ NYHA class II), unstable angina pectoris, or serious cardiac arrhythmia requiring medication.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening QTc interval > 480 msec will require investigator's evaluation on patient's eligibility. Subjects with left bundle branch block are excluded.
* Presence of a gastrointestinal condition that may affect drug absorption.
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2025-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Chheda, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Started | 24 | 27
Completed | 24 | 25
Not Completed | 0 | 2
Not completed — Did not start treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A: Retifanlimab+RT+Bevacizumab | Regimen B: Retifanlimab+RT+Bevacizumab+Epacadostat | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 81] | 58 [23 to 71] | 62 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 18 | 19 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) at 9 Months
Description: Overall survival is defined as the time interval from date of treatment start to date of a documented death event (death due to any cause) or date of censoring. If a patient has not had an event, OS will be censored at the date of last follow up.
Time Frame: At 9 months
Measure: Number (95% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
percentage of participants-Kaplan Meier | 67 [50 to 82] | 67 [51 to 89]

2. Primary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) at 12 Months
Description: as for outcome 1
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
percentage of participants-Kaplan Meier | 50 [34 to 75] | 38 [23 to 63]

3. Primary Outcome: Median Overall Survival (OS)
Description: as for outcome 1
Time Frame: Through 2 years after completion of treatment (estimated to be 4 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
months | 11.53 [9.79 to 17.97] | 10.55 [9.23 to 13.83]

4. Secondary Outcome: Change in Neurologic Functions as Measured by the Neurologic Function in Neuro-Oncology (NANO) Scale
Description: * There are 9 domains (gait, strength, ataxia, sensation, visual fields, facial strength, language, level of consciousness, and behavior).
  * Each domain is subdivided into 3 or 4 levels of function with scores based on discrete quantifiable measures. Each domain is scored from 0 to 3 points based on the severity of neurological deficit. A score of 0 indicates normal neurologic function, a score of 1 indicates mild impairment, 2 indicates severe impairment, and the highest score of 3 indicates the most severe level of deficit (incomplete hemianopsia) for that domain. Levels of function are distinguished by significant and measurable differences in order to avoid misinterpretation of subtle or nonspecific changes.
  * The total NANO score is the sum of the scores across all the 9 domains with a minimum score of 0 indicating normal function and a maximum score of 27 points indicating severe impairment. The total NANO score defines overall response criteria
Time Frame: Screening (mean 9 days, range 1-21 days prior to treatment) & at last assessment (31/49 patients measured at end of treatment, 18 patients' last measurement was on Cycle 2-23 with a mean of 5.8 cycles)
Population: Last assessment indicates the last time that a patient had an assessment of neurologic function measured via the NANO scale. Regimen A N=14 and Regimen B N=17 had the last assessment at end of treatment. Regimen A N=10 and Regimen B N=8 had the last assessment during treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
score on a scale
  Screening | 1.875 (2.071) | 2.12 (2.333)
  Last assessment | 2.952 (2.906) | 3.273 (2.865)

5. Secondary Outcome: Safety and Toxicity of Regimen as Measured by Immune Related Grade 3 or Higher Adverse Events Experienced by Participant
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting
Time Frame: 90 days after completion of treatment (estimated to be 2 years and 90 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
Participants
  Colitis | 1 | 0
  Diarrhea | 2 | 0
  Vomiting | 1 | 1
  Alanine aminotransferase increased | 2 | 1
  Aspartate aminotransferase increased | 0 | 1
  Seizure | 4 | 5
  Rash | 0 | 3

6. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) at 9 Months
Description: * Duration of time from start of treatment to radiographic progression or death due to any cause, whichever occurs first
  * Radiographic progression will be assessed using the RECIST 1.1. If the disease recurrence/progression assessment involves more than one date, the earliest date will be used as the event date. A patient will be censored at the date of the last radiographic disease assessment indicating a lack of disease progression, if any of the following occurs before documented disease progression: alive and lack evidence of progression at the end of study or at the time of analysis data cut-off, disease progression or death occurs right after missing data for a scheduled radiographic disease assessment, patient receives non-protocol treatment, or equivocal findings of recurrence - treatment may continue until the next scheduled assessment. If recurrence is confirmed at the next scheduled assessment, the date of recurrence should be the earlier date when recurrence was suspected
Time Frame: At 9 months
Measure: Number (95% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
percentage of participants-Kaplan Meier | 42 [26 to 67] | 21 [10 to 45]

7. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) at 12 Months
Description: as for outcome 6
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
percentage of participants-Kaplan Meier | 25 [13 to 50] | 4 [1 to 28]

8. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: as for outcome 6
Time Frame: Through 2 years after completion of treatment (estimated to be 4 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
Number analyzed (Participants) | 24 | 25
months | 6.98 [5.55 to 11.04] | 7.20 [5.78 to 8.61]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent through 90 days following the last date of treatment. All-cause mortality was collected from start of treatment through completion of follow-up (up to 4 years).
Arm/Group | Regimen A: Retifanlimab+RT+bevacizumab | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat
All-Cause Mortality (participants affected / at risk) | 24/24 | 24/25
Serious Adverse Events (participants affected / at risk) | 11/24 | 16/25
Other Adverse Events (participants affected / at risk) | 24/24 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Retifanlimab+RT+bevacizumab (N=24) | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Ehrlichhiosis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
BUN increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 0
Edema cerebral (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 2
Muscle weakness left-sided (Nervous system disorders) | 0 | 1
Muscle weakness right-sided (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 4 | 5
Stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 3
Psychosis (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Retifanlimab+RT+bevacizumab (N=24) | Regimen B: Retifanlimab+RT+bevacizumab+epacadostat (N=25)
Anemia (Blood and lymphatic system disorders) | 5 | 12
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2
Gum bleeding (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 3 | 6
Blurred vision (Eye disorders) | 1 | 1
Double vision (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 2
Eye stye (Eye disorders) | 1 | 0
Left homonymous hemianopsia (Eye disorders) | 0 | 1
Right homonymous hemianopsia (Eye disorders) | 0 | 1
Vision cut (Eye disorders) | 1 | 0
Vision decreased (Eye disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 7
Diarrhea (Gastrointestinal disorders) | 6 | 13
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 1
Mouth sore (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 12
Stomach pain (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 4 | 8
Chills (General disorders) | 3 | 1
Drooling (General disorders) | 1 | 0
Edema face (General disorders) | 3 | 2
Edema limbs (General disorders) | 3 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 14 | 15
Fever (General disorders) | 2 | 6
Flu like symptoms (General disorders) | 0 | 3
Gait disturbance (General disorders) | 3 | 2
Generalized edema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 0 | 3
Pain (fingers) (General disorders) | 1 | 0
Pain (foot) (General disorders) | 1 | 0
Pain (intermittent shooting pain) (General disorders) | 1 | 0
Pain (left hand pain) (General disorders) | 1 | 0
Pain (left hip, calf, and foot) (General disorders) | 1 | 0
Pain (shoulder) (General disorders) | 1 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 0 | 1
COVID-19 infection (Infections and infestations) | 3 | 3
Enterocolitis infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 2
Lip infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Thrush (Infections and infestations) | 2 | 2
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 2
Vaginal infection (Infections and infestations) | 0 | 1
Yeast infection on stomach (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 5
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 8
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 4
BUN increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 8
Decreased blood protein (Investigations) | 0 | 1
Hemoglobin increased (Investigations) | 2 | 2
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 15 | 15
Monocytes increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 4
Neutrophil count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 10 | 9
T4 increased (Investigations) | 0 | 1
Thyroid stimulating hormone increased (Investigations) | 6 | 3
Weight gain (Investigations) | 5 | 4
Weight loss (Investigations) | 9 | 10
White blood cell count increased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 10 | 6
Anorexia (Metabolism and nutrition disorders) | 5 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 12 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg and knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Anal cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 2 | 4
Concentration impairment (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 5
Dysarthria (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Dysphasia (Nervous system disorders) | 5 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 13
Hemineglect (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Left side neglect (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 3 | 3
Movements involuntary (Nervous system disorders) | 0 | 1
Muscle weakness left-sided (Nervous system disorders) | 0 | 5
Muscle weakness right-sided (Nervous system disorders) | 1 | 0
Occipital seizure (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 1
Phantom smells (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 3
Short-term memory loss (Nervous system disorders) | 0 | 1
Sour taste (Nervous system disorders) | 0 | 1
Spasticity (Nervous system disorders) | 0 | 1
Spinal stenosis (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 3 | 1
Word finding difficulties (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 2 | 2
Blunted affect (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 7 | 7
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 3
Hallucinations (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 5 | 3
Irritability (Psychiatric disorders) | 0 | 2
Glucosuria (Renal and urinary disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 2 | 4
Overactive bladder (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 13 | 14
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Amenorrhea (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Chafing (Skin and subcutaneous tissue disorders) | 1 | 0
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Facial cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Malar rash (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 11
Redness, small patch on right shoulder (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 17 | 16
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03532295/Prot_SAP_000.pdf